CLINICAL TRIAL: NCT01146301
Title: Does the Magnitude of Platelet Inhibition Inversely Correlate With the Number of TCD-detected Microemboli in Asymptomatic Patients Undergoing Carotid Artery Stenting Prior to Cardiac Surgery Who Are Being Pre-treated With 300 mg or 600 mg Loading Dose of Clopidogrel?
Brief Title: Platelet Inhibition and Transcranial Doppler (TCD)-Detected Microemboli During and After Carotid Artery Stenting (CAS) in Asymptomatic Patients Prior to Cardiac Surgery
Acronym: IMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Purpose: Treatment
Other Study IDs: R-06.44A
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Carotid Stenosis
Keywords: Platelet Aggregation Inhibitors; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Carotid Stenosis | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 300 mg Loading dose clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel
- 600 mg Loading dose of clopidogrel (Experimental)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — All patients will receive a loading dose of 600mg of study medication. The first group will receive 300 mg of clopidogrel and 300 mg placebo, the second group will receive 600mg of clopidogrel at least 24h before carotid stenting

SUMMARY:
As with coronary artery stenting, activation and embolisation of platelets occurs with carotid artery stenting (CAS). Based on promising data on the use of clopidogrel plus aspirin in coronary stenting this dual antiplatelet regimen has been introduced as adjunctive treatment during CAS. There is as yet, however, no randomized controlled trial which compared different loading doses of clopidogrel during CAS. Taking into account that a wide interindividual variability in the response to a loading of clopidogrel exists, this study is intended to establish the optimal loading dose of clopidogrel. Therefore platelet function testing and a 1-hour of postprocedural TCD (transcranial doppler) monitoring will be performed.

Objective: Firstly, to investigate whether the absolute magnitude of Platelet Inhibition inversely correlates with the number of TCD-detected microemboli during and after CAS in patients who are being pre-treated with either a 300 mg or a 600 mg loading dose of clopidogrel. Secondly, if there is any impact on early neurological outcome determined by the loading dose of clopidogrel.

DETAILED DESCRIPTION:
Carotid angioplasty with stent placement (CAS) has become a well-accepted treatment option for carotid artery stenosis. In combination with experience in CAS procedures and the introduction of protection devices and low-profile systems, the periprocedural risk of thromboembolic complications are comparable to that of standard surgical carotid endarterectomy (CEA) In our centre, all patients with severe asymptomatic carotid artery disease ( luminal diameter reduction of more than 80%, according to NASCET criteria) scheduled for cardiac surgery are eligible for CAS.

As with coronary artery stenting , activation and embolisation of platelets occurs with CAS. Based on promising data on the use of clopidogrel plus aspirin in coronary stenting, this dual antiplatelet regimen has been introduced in CAS. Specifically, an antiplatelet regimen with aspirin(300mg) and a 300 mg loading dose of clopidogrel at least 24 hours before carotid angioplasty has currently been the treatment of choice in carotid angioplasty with stent placement.

However, several studies have reported a wide interindividual variability in the response to a 300 mg loading of clopidogrel with a subsequent substantial proportion of patients not receiving the optimal benefit from it. Therefore, it has been suggested that a 600 mg loading dose will result in a faster onset, a higher responsiveness and a higher magnitude of platelet inhibition without any increase in bleeding complications. For these reasons, the interventional cardiology has already adopted the 600 mg loading dose regimen as standard of care during percutaneous coronary interventions. There is as yet, however, no randomized controlled trial which compared different loading doses of clopidogrel during CAS.

Using transcranial Doppler (TCD) monitoring of the middle cerebral artery during CAS, it is possible to register the number of TCD-detected microembolic signals during and after CAS. This monitoring enables the operator to diminish the risk of stroke during CAS. However, a significant number of patients develop an ischemic stroke in the hours following CAS after a symptom-free interval As published by van der Schaaf et al., in TCD monitoring after CEA, one hour of monitoring appeared to be effective to select those patients in whom the number of microemboli did not spontaneously decrease. More important, postoperative TCD monitoring was able to detect those patients who were at risk for new adverse cerebral events after the operation. Other studies demonstrate the potential application of ultrasonic emboli detection to examine the efficacy of new platelet agents in relatively small number of patients.

It remains to be established whether a higher magnitude of platelet inhibition before CAS has an additional protective effect by decreasing the microembolic load measured on TCD after the procedure. Moreover, such a TCD-monitoring post-CAS has not been performed systematically in the past and thus could reveal valuable information helpful to the understanding of post procedural cerebral complications and risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years of age
* patient accepted for CAS
* temporal window for TCD available

Exclusion Criteria:

* severe renal impairment (creatinine> 1.5mg/dl), abnormal liver function, malignancy, febrile disorder, acute or chronic inflammatory disease and other diseases influencing platelet reactivity
* extreme tortuositas or calcification of the lesion
* inadequate arterial access
* contraindication for angiography
* patient already receiving clopidogrel
* contra-indication to study drugs
* patients with active bleeding or at high-risk of bleeding
* uncontrolled hypertension ( > 180/110 mmHg) despite optimal medication
* pregnancy and women with inadequate anticonception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The number of TCD-detected microemboli during and immediately after the CAS procedure.
  The TCD monitoring of the Middle cerebral artery will be started during and immediately after the CAS procedure , using a 2 MHz TCD ultrasound probe. The Doppler spectra will be observed on-line and the audio-Doppler signal will be made audible in the angiography suite. For off-line analysis, the audio Doppler signals will be recorded on CD ROM. Analysis of recordings will be performed by an observer blinded to the clinical details and study group. Standard criteria for microemboli detection will be used.
The absolute level of platelet inhibition
  Blood samples for platelet function testing will be drawn at two different time-points: Before the administration of the study medication (baseline value) and immediately before the CAS-procedure. (time-interval will be approximately 24 hours) Platelet function testing will be performed with several platelet function assays: "classical"light transmittance aggregometry, The VerifyNow P2Y12 assay, Thrombelastograph® (TEG®) PlaletetMapping™ Assay and the Platelet function analyser (PFA-100).

SECONDARY OUTCOMES:
Periprocedural adverse cerebral events
  All patients will be assessed prior to treatment, at discharge and at 30 days following the procedure by an independent stroke neurologist. Strokes will be considered disabling (major), if patients has a modified Rankin score of more than 3, at 30 days after onset of symptoms. A minor stroke is defined as a Rankin score of 3 or less that resolves completely within 30 days. Transient ischemic attack and amaurosis fugax are diagnosed if the symptoms disappear within 24 hours. Fatal stroke is defined as death attributed to an ischemic or hemorrhagic stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- St-Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] Van Der Heyden J, Van Werkum J, Hackeng CM, Kelder JC, Breet NJ, Deneer VH, Ackerstaff RG, Tromp SC, De Vries JP, Vos JA, Suttorp MJ, Elsenberg EH, Van Neerven D, Schonewille WJ, Wolters F, Ten Berg JM. High versus standard clopidogrel loading in patients undergoing carotid artery stenting prior to cardiac surgery to assess the number of microemboli detected with transcranial Doppler: results of the randomized IMPACT trial. J Cardiovasc Surg (Torino). 2013 Jun;54(3):337-47. Epub 2012 Nov 8. PMID 23138609